CLINICAL TRIAL: NCT06510335
Title: Evaluation of a Lavender-based Natural Product System for Sleep Support
Brief Title: Lavender Essential Oil-based Product System for Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: dōTERRA International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DO-123048-SER
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: Lavender essential oil; Sleep quality; Gene expression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Masking Description: The study includes a single arm. Participants did not know the market name of the products they used. Products were packaged in plain bottles with the instruction label affixed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lavender essential oil-based product system (Experimental): Participants used the system in a sequential additive series. They used only the oil blend aromatically for 1 week, then the aromatic blend plus a topical stick application for 1 week, and then, for 4 weeks, the aromatic blend, the topical stick, and took 2 capsules of the dietary supplement nightly.
  Interventions: Other: Lavender essential oil-based product system

INTERVENTIONS:
Other: Lavender essential oil-based product system — Participants used the study products in a sequential, additive manner approximately 30-60 minutes before bedtime each night for 6 weeks. Usage consists of the following:
  * 20 drops of essential oil blend in approximately 250 mL of water in a diffuser, which operated for 8 hours at nighttime.
  * 3 x 6" swipes of the topical stick on the upper chest area, and 2 x 3" swipes on the inside of each wrist for topical application.
  * 2 capsules of the dietary supplement.
  Participants used the essential oil blend alone for 1 week, then added the topical stick for another 1 week. Finally, participants used the essential oil blend, the topical stick, and the dietary supplement for four weeks.
  Other Names: doTERRA Serenity Sleep System

SUMMARY:
The goal of this clinical trial is to learn whether lavender essential oil-based product system can affect gene expression, serum protein markers, and sleep quality in healthy volunteers. The main questions this study aims to answer are:

* Does the lavender essential oil-based product system affect gene expression and protein markers as measured in blood?
* Does the lavender essential oil-based product system affect subjective quality of life and sleep assessments?
* Is daily use of the product system safe, as measured by laboratory tests and adverse events?

The lavender essential oil-based product system contains three components: an essential oil blend, a topical stick, and a dietary supplement.

Participants will:

* Receive a fitness tracker to monitor their sleep and physical activity.
* Use the lavender essential oil-based product system for six weeks total according to this schedule:
* 1 week: Essential oil blend
* 1 week: Essential oil blend + topical stick
* 4 weeks: Essential oil blend + topical stick + dietary supplement
* Attend two study visits in which they provide blood and urine samples, and complete subjective sleep and quality of life assessments
* Complete weekly subjective sleep assessments from home

DETAILED DESCRIPTION:
This single-blind study will recruit healthy men and women to compare gene expression profile and serum protein markers before and after consumption of sleep system products for 6 weeks. Quality of life and sleep quality will be assessed using subjective surveys and questionnaires. Safety markers (liver and kidney function, hematology, urinalysis, and adverse events) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 35-50 years old
* Non-smokers
* Local to Pleasant Grove, Utah, and/or willing to come to clinical research center for study visits
* Willing and able to apply study products internally, topically and aromatically for about 6 weeks
* Willing to track use of study product on paper forms, via survey, or other means
* Willing to washout from all over-the-counter sleep aids, internally-consumed essential oils, alcohol, and lavender-based products for approximately 7 weeks
* Taking <100 mg caffeine daily, and willing to avoid consumption of caffeine after 3pm
* Not working night shift or swing shift
* Not consistently traveling to other time zones (or willing to arrange schedule to avoid during study)
* No known medical condition or sensitivity which would make the application of these study products unsafe
* Own a smart device that can download and run the accelerometer application
* Willing and able to keep the same sleeping arrangements as much as possible throughout the study
* Willing to receive and respond to regular texts, emails, and/or phone calls from study staff
* No pregnancy within the last 60 days or currently breastfeeding (females)
* Not currently or previously participating in any other clinical trial within the last 30 calendar days
* Signed informed consent, HIPAA Authorization, and Confidentiality Agreement
* No major medical conditions (especially cardiac, lung, metabolic, cancer, or sleep) under the active care of a doctor
* No prescription medications that may interfere with sleep (e.g. attention deficit hyperactivity disorder stimulants, antihistamines, psychiatric drugs, sleep medications, narcotics, etc.)
* No evidence of medical condition, significant disease or disorder, medication, or surgery within the past 12 months that may, in the judgment of the medical reviewer, put the participant at risk or affect study results, procedures, or outcomes (e.g. obstructive sleep apnea, morbid obesity, cardiometabolic disease, cancer, lung-related conditions)
* Willing and able (in the opinion of the investigator) to comply with all study requirements and procedures

Exclusion Criteria:

* Failure to meet any of the above inclusion criteria

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-11 (Actual)

PRIMARY OUTCOMES:
Gene expression | 6 weeks
  Gene expression analysis refers to a genome-wide quantification of methylation. This represents approximately 900,000 gene locations. The main feature performed is a differential methylation analysis to determine what has significantly changed from one time point to another.
Interleukin 6 (pg/mL) | 6 weeks
  Serum marker for inflammation
Cortisol (ug/mL) | 6 weeks
  Serum marker for stress response
Uric acid (mg/dL) | 6 weeks
  Serum marker for inflammation and signal of developing various disease processes
C-reactive protein (mg/L) | 6 weeks
  Serum marker for inflammation
Minutes awake | 6 weeks
  Mean nightly minutes awake determined by fitness tracker
Minutes asleep | 6 weeks
  Mean nightly minutes asleep determined by fitness tracker
Number of awakenings | 6 weeks
  Mean nightly number of awakenings determined by fitness tracker
Rapid Eye Movement (REM) sleep (minutes) | 6 weeks
  Mean nightly minutes of REM sleep determined by fitness tracker
Light sleep (minutes) | 6 weeks
  Mean nightly minutes of light sleep determined by fitness tracker
Deep sleep (minutes) | 6 weeks
  Mean nightly minutes of deep sleep determined by fitness tracker

SECONDARY OUTCOMES:
Albumin (g/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Blood urea nitrogen (BUN) (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Creatinine (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Alkaline phosphatase (U/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Alanine transaminase (ALT) (U/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Aspartate aminotransferase (AST) (U/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Calcium (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Carbon Dioxide (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Chloride (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Potassium (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Sodium (mmol/L) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Total bilirubin (mg/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Total protein (g/dL) | 6 weeks
  Item in comprehensive metabolic panel for safety assessment
Safety/tolerability | 6 weeks
  This study will monitor the occurrence and frequency of adverse events and safety through participant report and blood analyses.
Leeds Sleep Evaluation Questionnaire (LSEQ) | 6 weeks
  Validated, self-reported scale for the measurement of sleep quality. The LSEQ is a 10-item scale. Each item is scored 0 to 100. Higher scores indicate better sleep quality.
Short Form-20 (SF-20) scale | 6 weeks
  Validated, self-reported scale for the assessment of subjective quality of life. The SF-20 is a 20-item scale. Each item is scored 0-100. Higher scores indicate better subjective quality of life.
Functional Outcomes of Sleep Questionnaire (FOSQ) | 6 weeks
  Validated, self-reported scale for the measurement of sleep quality. The FOSQ is a 10-item scale. Higher scores indicate better sleep-related functional outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Stevens, PhD, Principal Investigator — doTERRA International
Locations (1):
- doTERRA International, Pleasant Grove, Utah, United States